CLINICAL TRIAL: NCT05697718
Title: A Phase I Study of Safety and Tolerability of Single-dose Human Umbilical Cord Mesenchymal Stem Cell (IxCell hUC-MSC-S) in Patients With Convalescent Phase of Ischemic Stroke
Brief Title: Clinical Trial of Human Umbilical Cord Mesenchymal Stem Cells (IxCell hUC-MSC-S) in the Treatment of Ischemic Stroke
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai IxCell Biotechnology Co., LTD (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LC-MSC-IS21004
Record Dates: First submitted 2022-12-27; First posted 2023-01-26 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group 1 (Experimental): Human umbilical cord mesenchymal stem cells（hMSCs）5.0×10^7 cells
  Interventions: Biological: MSC
- group 2 (Experimental): Human umbilical cord mesenchymal stem cells（hMSCs）10.0×10^7 cells
  Interventions: Biological: MSC
- group 3 (Experimental): Human umbilical cord mesenchymal stem cells（hMSCs）20.0×10^7 cells
  Interventions: Biological: MSC

INTERVENTIONS:
Biological: MSC — a single injection dose i.v.

SUMMARY:
To evaluate the safety and tolerability of IxCellhUC-MSC-S as a single intravenous infusion in convalescent patients with ischemic stroke.

To explore the efficacy of IxCellhUC-MSC-S as a single intravenous infusion in patients with convalescent ischemic stroke.

DETAILED DESCRIPTION:
MSCs are a type of stem cells derived from mesoderm with multidirectional differentiation potential. Studies have shown that MSCs have the potential to differentiate not only to bone, cartilage, fat and myogenic cells, but also to neurons.Among them, human cord blood mesenchymal stem cells are a kind of mature mesenchymal stem cells currently used. Human cord blood mesenchymal stem cells are ideal seed cells for tissue engineering. In addition to the advantages of convenient acquisition, rich source, easy expansion, etc., human cord blood collection also has the following advantages: (1) Collection of cord blood has no harm to maternal and newborn;(2) The cells are more primitive and have stronger ability of proliferation and differentiation;(3) Low immunogenicity, strong tolerance to human leukocyte antigen and low incidence of rejection;(4) The infection and transmission probability of tumor cells, viruses and pathogenic microorganisms is relatively low;(5) It does not involve many controversies in social, ethical and legal aspects.Current studies believe that the possible mechanisms of human umbilical cord mesenchymal stem cells in the treatment of stroke include replacing damaged nerve cells, promoting the proliferation and differentiation of endogenous nerve cells, secreting neurotrophic factors, promoting angiogenesis, reducing nerve cell apoptosis, and inhibiting inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 80 years old, both sexes;
2. Diagnosed with ischemic stroke of the anterior circulation at 12-24 weeks after the first stroke symptom onset (including W12 and W24);
3. National Institutes of Health Stroke Scale (NIHSS) score 6-20 points, and NlHSS score item 1a < 2 points;
4. Life expectancy ≥ 12 months;
5. Understand and comply with the study process, with informed consent form voluntarily signed by the patient or the authorized representatives.

Exclusion Criteria:

1. Current or previous epilepsy, dementia, Parkinson's disease, major depression, or other neurological disorders or mental illnesses that the investigator believes will affect their ability to participate in the study or affect the study evaluation;
2. Current or past intracranial hemorrhagic diseases (such as: cerebral hemorrhage, epidural hematoma, subdural hematoma, subarachnoid hemorrhage, ventricle hemorrhage, traumatic cerebral hemorrhage, etc.) or cerebral tumors, history of brain trauma, encephalitis and other symptoms leading to apoplexy;
3. Current or past severe cardiovascular disease；
4. Patients with pulmonary embolism, interstitial pneumonia, radiation pneumonia, drug-related pneumonia, severe impairment of lung function and other severe lung infections or other lung diseases (except those caused by stroke, bed rest after stroke or stroke treatment);
5. Have any other clinically serious medical conditions currently or in the past that the investigators judge unsuitable for inclusion in this study, including but not limited to severe liver (e.g., cirrhosis, etc.), kidney (e.g., kidney diseases requiring hemodialysis or peritoneal dialysis, etc.), blood (e.g., hemophilia with bleeding tendencies, etc.), endocrine (e.g.,Diabetes mellitus with difficult blood glucose control (blood glucose > 16.8mmol/L or < 2.8mmol/L), or complicated with severe neurovascular complications, etc.), immune system (active or uncontrolled autoimmune diseases, primary or secondary immune deficiencies, etc.), malignant tumors (except cured non-melanoma skin cancer, cervical or breast ductal carcinoma in situ), etc.;
6. Organ function level meet the following any one or more:

   absolute neutrophil cell count (ANC) < 1.5×109/L, platelet (PLT) < 100×109/L, hemoglobin (Hb) < 90g/L; Aspertate aminotransferase (AST) > 2.5×normal limit (ULN) and/or alanine aminotransferase (ALT) > 2.5×ULN, serum total bilirubin (TBIL) > 1.5×ULN; Creatinine (Cr) > 1.5×ULN; The international normalized ratio (INR) for those who did not receive anticoagulant or antithrombotic therapy > 1.7 or activated partial thromboplastin time (APTT) > 1.25×ULN, the international normalized ratio(INR) for those using anticoagulant or antithrombotic therapy > 3.0 or activated partial thromboplastin time (APTT) > 1.50×ULN.
7. Hepatitis B virus surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive for HBV-DNA, positive for hepatitis C virus antibody (HCVAb), treponema pallidum antibody (TPAb/RPR) or human immunodeficiency virus antibody (HIV), or within 14 days prior to receiving the test drug treatment,The emergence of any infected persons in need of systematic anti-infective treatment;
8. Allergic constitution or history, or allergic to the test drug or any component of the test drug;
9. Patients with MRI contraindications;
10. Positive blood pregnancy test results for female subjects of reproductive age within 7 days prior to receiving the experimental drug treatment;All women of reproductive age, fertile men or their spouses who refused to use appropriate contraception (including at least one barrier contraceptive) throughout the study period, and lactating women;
11. Those who required systemic corticosteroids (> 10mg/ day prednisone therapeutic dose) or other immunosuppressive agents within 14 days prior to receiving the trial drug or during the study period;
12. Patients who used butylphthalein within 3 weeks before receiving the experimental drug;
13. participated in any clinical trial and took any investigational drug within 3 months prior to receiving the investigational drug treatment (or the last time receiving the investigational drug did not exceed 5 half-lives, whichever is longer);
14. Patients who had severe trauma or major surgery within 3 months before receiving the experimental drug treatment, or who plan to undergo surgery during the trial period;Patients with a history of blood transfusion within 3 months before receiving the experimental drug treatment;
15. Those who had a history of drug abuse or alcoholism within 1 year before receiving the experimental drug treatment;
16. Those who have previously received other stem cell treatments;
17. Participants with other severe, acute, or chronic medical conditions that may increase the patient's risk or may interfere with the interpretation of the test results are judged by the investigator to be unsuitable for clinical trials.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-08-27 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 24 weeks
  Adverse events and serious adverse events
Laboratory test：blood routine | 24 weeks
Laboratory test：urine routine | 24 weeks
Laboratory test：blood biochemistry | 24 weeks
Laboratory test：coagulation function | 24 weeks
12-lead electrocardiogram | 24 weeks
Head magnetic resonance imaging（MRI） | 24weeks
Physical examination | 24weeks

SECONDARY OUTCOMES:
Preliminary efficacy | 24 weeks
  Changes in mRS scores at W12 and W24 compared to baseline after administration
Preliminary efficacy | 24 weeks
  The proportion of patients with a Barthel index (BI) score of ≥95 at W12 and W24 after administration
Preliminary efficacy | 24 weeks
  Changes in Barthel index (BI) at W12 and W24 compared to baseline after administration
Preliminary efficacy | 24 weeks
  Changes in the National Institutes of Health Stroke Scale (NIHSS) at W12 and W24 after administration compared to baseline
Preliminary efficacy | 24 weeks
  Changes in Fugl-Meyer（FM）scores at W12 and W24 compared to baseline after administration
Preliminary efficacy | 24 weeks
  Changes in infarct volume on MRI (FLAIR sequence) at W12 and W24 after administration compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: junwei Hao, Doctor, Principal Investigator — Xuanwu Hospital of Capital Medical University
Locations (2):
- China (2):
  - Xuanwu Hospital of Capital Medical University, Beijing, Beijing Municipality
  - Xuanwu Hospital of Capital Medical University, Beijing